CLINICAL TRIAL: NCT03095027
Title: Clinical Performance of a Silicone Hydrogel for Daily Disposable Wear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CLE383-C003
Record Dates: First submitted 2017-03-23; First posted 2017-03-29 (Actual); Results first posted 2019-02-04 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Refractive Error
Keywords: contact lens, silicone hydrogel, daily disposable, visual acuity
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Alcon Observer and Sponsor personnel were also masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- FID122819, then stenfilcon A (Other): FID122819 contact lenses worn first, followed by stenfilcon A contact lenses, as randomized. Each product worn in both eyes in a daily disposable mode for at least 8 hours per day, 5 days per week, for 1 week
  Interventions: Device: FID122819 contact lenses; Device: Stenfilcon A contact lenses
- Stenfilcon A, then FID122819 (Other): Stenfilcon A contact lenses worn first, followed by FID122819 contact lenses, as randomized. Each product worn in both eyes in a daily disposable mode for at least 8 hours per day, 5 days per week, for 1 week
  Interventions: Device: FID122819 contact lenses; Device: Stenfilcon A contact lenses

INTERVENTIONS:
Device: FID122819 contact lenses — Investigational spherical silicone hydrogel contact lenses for daily disposable wear
  Other Names: DDT2; Verofilcon A
Device: Stenfilcon A contact lenses — Commercially available spherical silicone hydrogel contact lenses for daily disposable wear
  Other Names: MyDay®

SUMMARY:
The purpose of this study is to compare the visual acuity of an investigational silicone hydrogel to a commercially available silicone hydrogel in contact lens wearers.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and sign an IRB-approved Informed Consent Form;
* Successful wear of spherical soft contact lenses in both eyes for a minimum of 5 days per week and 8 hours per day during the past 3 months:
* Manifest cylinder of ≤ 0.75 diopter (D) in each eye;
* Best corrected visual acuity (BCVA) of 20/25 or better in each eye;
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Any anterior segment infection, inflammation, abnormality or disease (including systemic) that contraindicates contact lens wear, as determined by the Investigator;
* Any use of systemic or ocular medications for which contact lens wear could be contraindicated, as determined by the Investigator;
* History of refractive surgery or plan to have refractive surgery during the study;
* Ocular or intraocular surgery within the previous 12 months or planned during the study;
* Current or history of pathologically dry eye in either eye that, in the opinion of the Investigator, would preclude contact lens wear;
* Any previous or current wear of MYDAY;
* Habitually wearing monovision or multifocal lenses during the last 3 months;
* Routinely sleeping in lenses for at least 1 night per week over the last 3 months prior to enrollment;
* Any use of topical ocular medications and artificial tear or rewetting drops that would require instillation during contact lens wear;
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-04-19 (Actual); Primary Completion 2017-05-15 (Actual); Study Completion 2017-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Clinical Manager, Trial Management Operations, Study Director — Alcon, A Novartis Division
Locations (3):
- United States (3):
  - Alcon Investigative Site, Longwood, Florida
  - Alcon Investigative Site, Maitland, Florida
  - Alcon Investigative Site, Johns Creek, Georgia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 3 study centers located in the United States.
Pre-assignment Details: Of the 54 enrolled, 3 subjects were exited as screen failures prior to randomization. This reporting group includes all randomized subjects (51).
Period: Period 1, First Week of Wear
Arm/Group | FID122819, Then Stenfilcon A | Stenfilcon A, Then FID122819
Started (As Treated; 1 subject randomized to stenfilcon A/FID122819 exposed to FID122819/stenfilcon A instead) | 27 | 24
Completed | 27 | 24
Not Completed | 0 | 0
Period: Period 2, Second Week of Wear
Arm/Group | FID122819, Then Stenfilcon A | Stenfilcon A, Then FID122819
Started | 27 | 24
Completed | 26 | 24
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all randomized subjects exposed to any study lens evaluated in this study. Each subject/eye was analyzed according to the respective randomized lens, irrespective of the exposure (Full Analysis Set).
Groups:
- Overall: FID122819 and stenfilcon A contact lenses worn during Period 1 and Period 2 in a crossover assignment.
Arm/Group | Overall
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.5 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 49
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity (VA)
Description: VA was assessed and collected using a Snellen chart. Conversion to logMAR (logarithm of the minimum angle of resolution) was performed. A logMAR acuity of 0.0 corresponds to 20/20 Snellen acuity, with a negative value denoting better than 20/20 visual acuity. Both eyes contributed to the analysis.
Time Frame: Baseline/Dispense (Day 1), Week 1, each product
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: Eyes
Groups:
- FID112819: FID122819 contact lenses worn during Period 1 or Period 2 for 1 week
- Stenfilcon A: Stenfilcon A contact lenses worn during Period 1 or Period 2 for 1 week
Arm/Group | FID112819 | Stenfilcon A
Number analyzed (Participants) | 51 | 51
Number analyzed (Eyes) | 102 | 102
logMAR
  Dispense | -0.08 (0.06) | -0.09 (0.06)
  Week 1: number analyzed (Participants) | 51 | 50
  Week 1: number analyzed (Eyes) | 102 | 100
  Week 1 | -0.09 (0.06) | -0.09 (0.06)
Statistical Analysis 1: Comparison: FID112819 vs Stenfilcon A; Test type: Non-Inferiority — The pre-specified non-inferiority margin is 0.05. With a sample size of 10, there was approximately 80% power to reject the null hypothesis of inferiority in visual acuity with assumed standard deviation of 0.0474 (one-sided alpha=0.05); LSM Difference = 0.00, 95% CI 1-sided [upper limit 0.01], Standard Error of Mean 0.00

ADVERSE EVENTS:
Time Frame: Dispense through study completion, an average of 2 weeks
Description: Adverse Events (AEs) were any untoward medical occurrence, unintended disease or injury, or untoward clinical signs in subjects, users or other persons, whether or not related to the investigational medical device. AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator. This analysis population includes all subjects/eyes exposed to any study lens evaluated (Safety Analysis Set), based on treatment-specific exposure.
Groups:
- FID122819: Subjects exposed to FID122819 contact lenses during Period 1 or Period 2
- Stenfilcon A: Subjects exposed to stenfilcon A contact lenses during Period 1 or Period 2
Arm/Group | FID122819 | Stenfilcon A
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/51
Other Adverse Events (participants affected / at risk) | 0/51 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2017-03-07): https://cdn.clinicaltrials.gov/large-docs/27/NCT03095027/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-21): https://cdn.clinicaltrials.gov/large-docs/27/NCT03095027/SAP_001.pdf